CLINICAL TRIAL: NCT03839394
Title: A Clinic-Based Case Manager Administered Telephone Intervention to Reduce Cardiovascular Disease Risk in Persons Living With HIV
Brief Title: Case Managers for CVD Risk Reduction in HIV Clinic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00085562; K23HL137611-01A1 (NIH)
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Disease; HIV
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational pamphlets + telephone (Experimental)
  Interventions: Behavioral: Telephone; Other: Educational pamphlets
- Educational pamphlets (Active Comparator)
  Interventions: Other: Educational pamphlets

INTERVENTIONS:
Behavioral: Telephone — A series of educational pamphlets on CVD risk reduction plus a telephone-based CVD risk reduction curriculum will be administered by Clinic-Based Case Managers (CCMs). Six modules will be given over 24 weeks in a rotating fashion on topics relevant to CVD risk. Subjects will be given the pamphlets every 2 weeks corresponding with the first time they receive the telephone - based module.
  Arms: Educational pamphlets + telephone
Other: Educational pamphlets — A series of 6 handouts will be given to controls once monthly over 6 months on the same topics presented in the telephone modules. Educational packets will be primarily drawn from free printed material available at www.learningaboutdiabetes.org and the American Heart Association website.

SUMMARY:
The purpose of the study is to assess the efficacy of a case manager/social worker administered, telephone-based educational curriculum in improving cardiovascular disease related outcomes among HIV-infected clinic patients.

DETAILED DESCRIPTION:
Fifty high Cardiovascular Disease Risk (CVD) risk clinic patients will be randomized 1:1 to receive either a series of educational pamphlets on CVD risk reduction plus a telephone-based CVD risk reduction curriculum delivered over 24 weeks [intervention arm], or the educational pamphlets alone [control arm]. Anthropomorphic data, blood pressure and lipid profiles will be obtained from patients to assess the efficacy of the intervention in reducing blood pressure and serum low-density lipoprotein levels (LDL).

ELIGIBILITY:
Inclusion Criteria:

* In care at the Duke Infectious Diseases Clinic for HIV and for at least 24 months
* On antiretroviral therapy
* 2013 American Heart Association 10-year ASCVD risk score ≥ 15%, with a diagnosis of either hypertension or hyperlipidemia
* English literate (able to speak and read at a 6th grade level)
* Subjects must have the capacity to give legally effective consent.

Exclusion Criteria:

* Patients with prior diagnosis of acute coronary syndrome, stroke, peripheral vascular disease, and end stage renal disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nwora L Okeke, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website referring to educational materials to be shared as part of this intervention — http://www.learningaboutdiabetes.org
- See also: Website referring to educational materials to be shared as part of this intervention — https://www.heart.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Started | 25 | 24
Completed | 19 | 14
Not Completed | 6 | 10
Not completed — Lost to Follow-up | 6 | 8
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (6.1) | 54.0 (9.4) | 56.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 24 | 23 | 47
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 15 | 35
  White | 4 | 7 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Ambulatory Systolic Blood Pressure
Description: Change of systolic blood pressure will be assessed as an absolute continuous variable, and as a proportion or persons who achieve >5mmHg reduction in systolic blood pressure from baseline. Reported here is the change from baseline to 72 weeks.
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Number analyzed (Participants) | 19 | 14
mmHg | 1.9 (15.0) | -10.7 (10.9)
Statistical Analysis 1: Comparison: Educational Pamphlets + Telephone vs Educational Pamphlets; This was a pilot study positioned to determine the effect size of a clinic-based intervention that has not been evaluated previously. Therefore, sample size was determined to be adequate to discern an effect size, but not powered to determine definitive statistical significance; Test type: Other; p = 0.012, t-test, 2 sided

2. Primary Outcome: Number of Participants Who Achieve >5mmHg Reduction in Systolic Blood Pressure From Baseline
Time Frame: Baseline, 72 weeks
Population: Participants with data collected at both timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Number analyzed (Participants) | 19 | 14
Participants | 7 | 10
Statistical Analysis 1: Comparison: Educational Pamphlets + Telephone vs Educational Pamphlets; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.05, Z-test of Proportions

3. Primary Outcome: Change in Non-HDL (High Density Lipoprotein Cholesterol) Levels
Description: Assessment of the absolute change in fasting calculated non-high density lipoprotein cholesterol over the study period. Reported here is the change from baseline to 72 weeks.
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Number analyzed (Participants) | 16 | 15
mg/dL | -5.7 (36.2) | -1.5 (37.4)
Statistical Analysis 1: Comparison: Educational Pamphlets + Telephone vs Educational Pamphlets; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.750, t-test, 2 sided

4. Secondary Outcome: Total Change in Body Weight
Description: Total change in body weight from baseline over the study period. Reported here is the change from baseline to 72 weeks.
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Number analyzed (Participants) | 19 | 14
kg | -1.8 (5.1) | -2.1 (4.8)
Statistical Analysis 1: Comparison: Educational Pamphlets + Telephone vs Educational Pamphlets; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.860, t-test, 2 sided

5. Secondary Outcome: Change in 10-year Atherosclerotic Cardiovascular Disease (ASCVD) Risk Score
Description: The global cardiovascular disease risk as calculated by the American College of Cardiology/American Heart Association's 10-year risk calculator. The ASCVD risk score is a calculation of the 10-year risk of having a cardiovascular problem, such as a heart attack or stroke. The ASCVD risk score is given as a percentage, which represents the chance of having heart disease or stroke in the next 10 years. 0 to 4.9 = low risk, 5 to 7.4 = borderline risk, 7.5 to 20 = intermediate risk, >20 = high risk. Reported here is the change from baseline to 72 weeks.
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks
Population: Participants with data collected at both timepoints.
Measure: Mean (Standard Deviation); unit: percentage of risk
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
Number analyzed (Participants) | 12 | 6
percentage of risk | -1.0 (4.1) | -0.4 (3.3)
Statistical Analysis 1: Comparison: Educational Pamphlets + Telephone vs Educational Pamphlets; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.760, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Description: All significant medical events reported in all participants during the study observation period were abstracted from the clinical record, recorded in the study record and adjudicated for association with study intervention by the study PI.
Arm/Group | Educational Pamphlets + Telephone | Educational Pamphlets
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/25 | 3/24
Other Adverse Events (participants affected / at risk) | 9/25 | 3/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Educational Pamphlets + Telephone (N=25) | Educational Pamphlets (N=24)
incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1
deep venous thrombosis (Blood and lymphatic system disorders) | 0 | 1
epididimytis (Reproductive system and breast disorders) | 0 | 1
stroke (Nervous system disorders) | 1 | 0
suicidal ideation (Psychiatric disorders) | 1 | 0
auditory hallucinations (Psychiatric disorders) | 1 | 0
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
gastroenteritis (Gastrointestinal disorders) | 1 | 0
colonic polyps (Gastrointestinal disorders) | 1 | 0
esophageal mass (Gastrointestinal disorders) | 1 | 0
syncope (Cardiac disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Educational Pamphlets + Telephone (N=25) | Educational Pamphlets (N=24)
cataract surgery (Surgical and medical procedures) | 0 | 1
assault (Social circumstances) | 0 | 1
anal condyloma (Gastrointestinal disorders) | 0 | 1
colonoscopy (Surgical and medical procedures) | 2 | 0
direct laryngoscopy (Surgical and medical procedures) | 1 | 0
upper endoscopy (Surgical and medical procedures) | 1 | 0
laryngeal mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hip replacement (Surgical and medical procedures) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0
gonorrhea (Infections and infestations) | 1 | 0
scapular abscess (Infections and infestations) | 1 | 0
transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
inguinal hernia (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT03839394/Prot_SAP_001.pdf
  • Informed Consent Form (2021-06-29): https://cdn.clinicaltrials.gov/large-docs/94/NCT03839394/ICF_000.pdf